CLINICAL TRIAL: NCT03606343
Title: Teaching Academic Success Skills to Middle School Students With Autism Spectrum Disorders (ASD) With Executive Functioning Deficits - in Clinical Setting
Brief Title: Teaching Academic Success Skills to Students With Autism Spectrum Disorders in Clinical Setting
Acronym: TASK-R21
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R21HD090334-01A1 (NIH)
Record Dates: First submitted 2018-05-16; First posted 2018-07-30 (Actual); Results first posted 2020-11-24 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-11

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Open trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open Trial (Experimental): Group based treatment targeting academic executive functioning skills such as organization, planning, and study skills. Likely to be 7 90-minute sessions attended weekly by parents and teens
  Interventions: Behavioral: Teaching Academic Skills to Kids

INTERVENTIONS:
Behavioral: Teaching Academic Skills to Kids — Group treatment

SUMMARY:
The goal of the study is to develop an academic EF intervention, Teaching Academic Skills to Kids (TASK), for high functioning (i.e., IQ score ≥80) middle-school youth with ASD and EF deficits.

Aim 1: Use focus group methodology and advice from expert consultants to develop the TASK intervention targeting academic EF skills for middle school youth with ASD that is tailored to the unique needs of these individuals (e.g., content specific to ASD EF deficits, incorporate evidence-based teaching principles and methods for ASD).

Aim 2: Examine the feasibility and acceptability of TASK in 3 open trials to assess initial feasibility and efficacy.

DETAILED DESCRIPTION:
The goal of the study is to develop an academic EF intervention, Teaching Academic Skills to Kids (TASK), for high functioning (i.e., IQ score ≥80) middle-school youth with ASD and EF deficits.

Aim 1: Develop the TASK intervention targeting academic EF skills for middle school youth with ASD that is tailored to the unique needs of these individuals (e.g., content specific to ASD EF deficits, incorporate evidence-based teaching principles and methods for ASD). A methodologically rigorous, well-integrated iterative and collaborative design process with input from multiple stakeholders, including school mental health professionals, teachers, parents, and youth with ASD, will be utilized.

Aim 2: Examine the feasibility and acceptability of TASK in 3 open trials including the feasibility of: 1) implementing the measurement protocol, 2) operationalizing intervention delivery, 3) assessing both trained and untrained areas of functioning, 4) assessing whether improvements in academic EF skills (proposed mechanism of treatment) are related to functional educational outcomes (e.g., homework behaviors, grades), and 5) exploring the data for potential treatment moderators (e.g., gender, severity). It is hypothesized that TASK will be feasible, acceptable (attendance, satisfaction), and will result in improved academic EF skills associated with reduced academic impairment and homework problems.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autism spectrum disorder
* IQ >80
* 7th grade at time of intervention
* mainstreamed classroom
* executive functioning problems identified on parent or teacher BRIEF-2

Exclusion Criteria:

* danger to self or others

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with other researchers via the National Database for Autism Research (NDAR) without exposing personally identifiable information.
Supporting Information: Study Protocol
Time Frame: after August 31, 2019 when study is completed, indefinitely available.
Access Criteria: specified by NDAR
URL: http://ndar.nih.gov

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Youth with ASD without ID attending middle school and their parents were recruited in the 2018-2019 academic school year via letters, flyers, and emails targeted at individuals who had received services at a hospital outpatient clinic specializing in assessment and treatment of autism.
Period: Overall Study
Arm/Group | Open Trial
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Middle school student with Autism Spectrum Disorder without Intellectual Disability
Arm/Group | Open Trial
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.2 (1.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21
Kauffman Brief Intelligence Test - Second Edition [Mean (Standard Deviation); unit: scores on a scale] — This is a brief IQ test. The Standard Score has a mean of 100 and a standard deviation of 15. Higher scores indicate higher intelligence. The range of possible scores is 40 to 160
  scores on a scale | 109.7 (13.8)

OUTCOME MEASURES:

1. Primary Outcome: Children's Organizational Skills Scale
Description: The Children's Organizational Skills Scale is a rating scale of organization and executive functioning. A T-score is reported. A T-score of 50 indicates the population mean with a standard deviation of 10. Range of possible T-scores is 40 to 90. Higher T-scores indicate poorer organization/executive functioning. We present baseline (before intervention) and 3 month outcome (post intervention) T-scores as rated by the parent.
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Open Trial
Number analyzed (Participants) | 21
T-Score
  Baseline Parent Total COSS T-Score | 66.14 (9.43)
  3 months Parent Total COSS T-Score | 57.24 (9.96)

2. Primary Outcome: Behavior Rating Inventory of Executive Function - Second Edition
Description: The Behavior Rating Inventory of Executive Function - Second Edition is a parent rating scale of executive functioning. A T-score is reported. A T-score of 50 indicates the population mean with a standard deviation of 10. Range of possible T-scores is 40 to 90. Higher T-scores indicate poorer executive functioning. We present baseline (before intervention) and 3 month outcome (post intervention) T-scores.
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Open Trial
Number analyzed (Participants) | 21
T-score
  Baseline Parent General Executive Composite T-Scor | 71.86 (8.62)
  3 month Parent General Executive Composite T-Scor | 66.57 (8.78)

3. Primary Outcome: Homework Problem Checklist
Description: The Homework Problem Checklist is a rating scale of homework behavior completed by the parent. There are two subscales generated: Homework Completion Behaviors & Homework Management Behaviors. Scale is rated on a 0 = never to 3 = very often scale and a sum of scores is computed for each subscale. Range of scores for Homework Completion Behaviors is 0 to 36. Range of scores for Homework Management Behaviors is 0 to 21. We present baseline (before intervention) and 3 month outcome (post intervention) scores for each subscale. Higher scores indicate worse outcome.
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Trial
Number analyzed (Participants) | 21
score on a scale
  Baseline Homework Completion Behaviors | 24.24 (6.58)
  3 Month Homework Completion Behaviors | 15.71 (7.63)
  Baseline Homework Management Behaviors | 8.33 (6.09)
  3 Month Homework Management Behaviors | 4.57 (4.40)

4. Secondary Outcome: Woodcock Johnson Tests of Achievement - Third Edition Basic Writing Subtest
Description: The Woodcock Johnson is an academic performance measure administered to the child. A standard score of 100 indicates the population mean with a standard deviation of 15 (range of 40 to 170). Lower standard scores are worse. We present baseline (before intervention) and 3 month outcome (post intervention) for the Basic Writing subtest.
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Trial
Number analyzed (Participants) | 21
score on a scale
  Baseline WJ-III Basic Writing | 103.85 (11.91)
  3 Month WJ-III Basic Writing | 105.80 (13.51)

5. Secondary Outcome: Classroom Performance Survey
Description: The Classroom Performance Survey is a teacher rating scale of classroom behavior. The scale is rated 1 = always to 5 = never. An academic competence mean score is computed (range 1 to 5) with higher scores indicating a worse outcome. We present baseline (before intervention) and 3 month outcome (post intervention) total mean score.
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Trial
Number analyzed (Participants) | 21
score on a scale
  Baseline Academic Competence | 2.02 (.95)
  3 Month Academic Competence | 1.91 (0.93)

6. Secondary Outcome: Academic Performance Rating System
Description: The Academic Performance Rating System is a teacher rating scale of academic performance. Items are rated 1 = Never to 5 = Very often and the items are summed to generate a Total Score (range 19 to 95) with higher scores worse indicating a worse outcome. We present the Total score at baseline (before intervention) and 3 month outcome (post intervention).
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Trial
Number analyzed (Participants) | 21
score on a scale
  Baseline APRS Total | 45.83 (12.14)
  3 Month APRS Total | 52.11 (14.58)

7. Secondary Outcome: Parenting Relationship Questionnaire - Communication Subscale
Description: The Parenting Relationship Questionnaire is completed by parents to describe their parenting relationship with the teen. A T-score is reported for the Communication subscale. A T-score of 50 indicates the population mean with a standard deviation of 10. Range of possible T-scores is 40 to 90. Lower T-scores indicate poorer communication. We present baseline (before intervention) and 3 month outcome (post intervention) T-scores.
Time Frame: baseline, 3 months
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Open Trial
Number analyzed (Participants) | 21
T-Score
  Baseline Communication T-Score | 41.1 (8.7)
  3 Month Communication T-Score | 43.2 (8.3)

ADVERSE EVENTS:
Time Frame: 3 months
Description: Adverse event monitoring occurred at each assessment visit. Participants were asked if they have had any adverse experiences since the last visit.
Arm/Group | Open Trial
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-22): https://cdn.clinicaltrials.gov/large-docs/43/NCT03606343/Prot_SAP_000.pdf